CLINICAL TRIAL: NCT00401544
Title: Once Per Cycle Treatment of Anemia With Darbepoetin Alfa With Iron in Subjects With Non Myeloid Malignancies
Brief Title: Darbepoetin Alfa With or Without Intravenous (IV) Iron
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060103
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Anemia; Non-Myeloid Malignancies
Keywords: anemia; chemotherapy induced anemia; darbepoetin alfa; cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa; Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Darbepoetin alfa 300 μg plus IV Iron (Experimental): Darbepoetin alfa 300 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
  Interventions: Drug: darbepoetin alfa; Drug: IV iron dextran
- Darbepoetin alfa 300 μg (Experimental): Darbepoetin alfa 300 μg subcutaneous injection every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
  Interventions: Drug: darbepoetin alfa
- Darbepoetin alfa 500 μg (Experimental): Darbepoetin alfa 500 μg subcutaneous injection every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
  Interventions: Drug: darbepoetin alfa
- Darbepoetin alfa 500 μg plus IV Iron (Active Comparator): Darbepoetin alfa 500 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
  Interventions: Drug: darbepoetin alfa; Drug: IV iron dextran

INTERVENTIONS:
Drug: darbepoetin alfa — Darbepoetin alfa administered by subcutaneous injection.
  Other Names: Aranesp®
Drug: IV iron dextran — Administered by intravenous (IV) injection.
  Other Names: INFeD®; Cosmofer®
  Arms: Darbepoetin alfa 300 μg plus IV Iron; Darbepoetin alfa 500 μg plus IV Iron

SUMMARY:
To deterime the efficacy of 500 μg and 300 μg darbepoetin alfa administered subcutaneously (SC) on an every 3 weeks (Q3W) schedule, and the effect of intravenous (IV) iron supplementation in the treatment of anemia in patients with non-myeloid malignancies who were receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Active non myeloid malignancy(cies) including lymphocytic leukemias
* Received chemotherapy and expected to receive at least 8 additional weeks of cyclic cytotoxic chemotherapy
* Anemia due to chemotherapy (screening Hgb <or = 10.0 g/dL)
* at least 18 years of age at screening

Exclusion Criteria:

* Acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML), or myelodysplastic syndromes (MDS)
* Other underlying hematologic disorder, which could cause anemia, other than a non myeloid malignancy
* Active bleeding
* Severe, unstable, active chronic inflammatory disease (eg ulcerative disease, peptic ulcer disease, rheumatoid arthritis)
* Active, unstable systemic or chronic infection
* Planned elective surgery during the study where significant blood loss is expected
* Unstable angina, or uncontrolled cardiac arrhythmia
* Uncontrolled hypertension (diastolic blood pressure > 100 mmHg)
* History of pure red cell aplasia (PRCA)
* History of deep venous thrombosis
* Known positive human immunodeficiency virus (HIV) test or acquired immune deficiency syndrome (AIDS) status
* Any red-blood-cell (RBC) transfusion within 28 days before randomization and/or during screening
* Currently receiving thalidomide or lenalidomide without prophylactic anticoagulant therapy
* Currently receiving or planned to receive myeloablative radiation therapy
* Received bone marrow or stem cell transplant in the 6 months prior to screening or planned during the study
* Received any erythropoietic therapy within 28 days before randomization and/or during screening (eg rHuEPO or darbepoetin alfa)
* Known sensitivity to any erythropoietic agents, the investigational product or its excipients to be administered during this study
* Known sensitivity to iron administration
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Auerbach M, Silberstein PT, Webb RT, Averyanova S, Ciuleanu TE, Shao J, Bridges K. Darbepoetin alfa 300 or 500 mug once every 3 weeks with or without intravenous iron in patients with chemotherapy-induced anemia. Am J Hematol. 2010 Sep;85(9):655-63. doi: 10.1002/ajh.21779. PMID 20661916
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 18 December 2006 through 27 August 2007.
Pre-assignment Details: A total of 243 patients were randomizd and 238 received study drug (4 participants in the Darbepoetin alfa 300 μg plus Iron group and 1 in the Darbepoetin alfa 500 μg plus Iron group were not treated)
Groups:
- Darbepoetin Alfa 300 μg Plus Iron: Darbepoetin alfa 300 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
- Darbepoetin Alfa 500 μg Plus Iron: Darbepoetin alfa 500 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
Period: Overall Study
Arm/Group | Darbepoetin Alfa 300 μg Plus Iron | Darbepoetin Alfa 300 μg | Darbepoetin Alfa 500 μg Plus Iron | Darbepoetin Alfa 500 μg
Started | 56 (Randomized and treated) | 62 (Randomized and treated) | 60 (Randomized and treated) | 60 (Randomized and treated)
Completed | 38 | 44 | 48 | 44
Not Completed | 18 | 18 | 12 | 16
Not completed — Adverse Event | 5 | 1 | 1 | 1
Not completed — Death | 3 | 6 | 2 | 5
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 6 | 5
Not completed — Physician Decision | 1 | 3 | 0 | 0
Not completed — Ineligibility determined | 0 | 1 | 0 | 2
Not completed — Disease progression | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa 300 μg Plus Iron | Darbepoetin Alfa 300 μg | Darbepoetin Alfa 500 μg | Darbepoetin Alfa 500 μg Plus Iron | Total
Number analyzed (Participants) | 56 | 62 | 60 | 60 | 238
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (12.5) | 62.1 (14.1) | 66.7 (12.0) | 62.3 (13.3) | 63.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 44 | 33 | 47 | 158
  Male | 22 | 18 | 27 | 13 | 80
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 7 | 5 | 9 | 11 | 32
  Hispanic or Latino | 2 | 7 | 1 | 3 | 13
  Asian | 2 | 1 | 0 | 0 | 3
  Other | 0 | 1 | 0 | 0 | 1
  White or Caucasian | 45 | 48 | 50 | 46 | 189
FACT-Fatigue Score [Mean (Standard Deviation); unit: Units on a scale] — Functional Assessment of Cancer Therapy (FACT) - Fatigue subscale score, ranging from 0 to 52, where 0 = worst outcome and higher scores represent less fatigue.
  Units on a scale | 28.54 (12.32) | 30.24 (12.46) | 28.60 (11.95) | 30.25 (11.79) | 29.44 (12.08)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 9.4 (1.1) | 9.4 (0.9) | 9.4 (1.2) | 9.2 (0.9) | 9.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved the Target Hemoglobin Level, by Darbepoetin Alfa Dose
Description: Target hemoglobin was defined as ≥ 11 g/dL during the treatment period in the absence of a red blood cell (RBC) transfusion on the day of measurement or during the preceding 28 days.
Time Frame: From Week 1 to Week 16
Population: Subset of Primary Analysis Set, composed of all randomized participants who received at least one dose of blinded study medication, who had baseline hemoglobin values < 11.0 g/dL.
Measure: Number; unit: Participants
Groups:
- Combined Darbepoetin Alfa 300 μg: Darbepoetin alfa 300 μg subcutaneous injection with or without intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
- Combined Darbepoetin Alfa 500 μg: Darbepoetin alfa 500 μg subcutaneous injection with or without intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
Arm/Group | Combined Darbepoetin Alfa 300 μg | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 112 | 115
Participants | 71 | 82
Statistical Analysis 1: Comparison: Combined Darbepoetin Alfa 500 μg; Test type: Superiority or Other; Percentage of participants = 71, 95% CI [63 to 80] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Combined Darbepoetin Alfa 300 μg; Test type: Superiority or Other; Percentage of participants = 63, 95% CI [54 to 72] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

2. Primary Outcome: Number of Participants Who Achieved the Target Hemoglobin Levels, by IV Iron Usage
Description: as for outcome 1
Time Frame: From Week 1 to Week 16
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Combined Without Iron Groups: Darbepoetin alfa 300 μg or 500 μg subcutaneous injection every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
- Combined With Iron Groups: Darbepoetin alfa 300 μg or 500 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 117 | 110
Participants | 73 | 80
Statistical Analysis 1: Comparison: Combined With Iron Groups; Test type: Superiority or Other; Percentage of participants = 73, 95% CI [64 to 81] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Combined Without Iron Groups; Test type: Superiority or Other; Percentage of participants = 62, 95% CI [54 to 71] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

3. Secondary Outcome: Time to Achieve Target Hemoglobin Level, by Darbepoetin Alfa Dose
Description: The time to target hemoglobin is the interval in weeks between study day 1 and the first day that a hemoglobin value ≥ 11.0 g/dL is observed during the treatment period. If a participant did not achieve the target hemoglobin by the time of withdrawal or the end of the treatment period (EOTP), the time to target hemoglobin was censored on the day of the last hemoglobin measurement or the EOTP, whichever was earlier. Median was calculated using Kaplan-Meier estimates.
Time Frame: From Week 1 to Week 16
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Combined Darbepoetin Alfa 300 μg | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 112 | 115
Weeks | 10.0 [7.0 to 11.0] | 8.0 [6.0 to 10.0]

4. Secondary Outcome: Time to Achieve the Target Hemoglobin Level, by IV Iron Usage
Description: as for outcome 3
Time Frame: From Week 1 to Week 16
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 117 | 110
Weeks | 9.0 [7.0 to 11.0] | 8.0 [5.0 to 10.0]

5. Secondary Outcome: Change From Baseline in Hemoglobin Concentration, by Darbepoetin Alfa Dose
Description: Change in hemoglobin concentration from Baseline to the end of the treatment period (Week 16).
Time Frame: Baseline and Week 16
Population: Primary Analysis Set, composed of all participants who were randomized, properly consented, and received at least one dose of blinded study drug. Imputation by last value carried forward (LVCF) was applied.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Combined Darbepoetin Alfa 300 μg | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 118 | 120
g/dL | 1.5 (1.8) | 1.6 (1.8)

6. Secondary Outcome: Change From Baseline in Hemoglobin Concentration, by IV Iron Usage
Description: Change in hemoglobin concentration from Baseline to the end of the treatment period (Week 16).
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 122 | 116
g/dL | 1.3 (1.7) | 1.9 (1.8)

7. Secondary Outcome: Number of Participants With ≥ 1 Red Blood Cell Transfusion From Week 1 to End of Study, by Darbepoetin Alfa Dose
Description: The number of participants with ≥ 1 red blood cell (RBC) transfusion from week 1 to end of study (EOS). Participants with a hemoglobin value ≤ 8 g/dL but no RBC transfusion were counted as having had a transfusion.
Time Frame: From Week 1 to Week 16
Population: Primary Analysis Set, composed of all participants who were randomized, properly consented, and received at least one dose of blinded study drug.
Measure: Number; unit: Participants
Arm/Group | Combined Darbepoetin Alfa 300 μg | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 118 | 120
Participants | 45 | 43
Statistical Analysis 1: Comparison: Combined Darbepoetin Alfa 500 μg; Test type: Superiority or Other; Percentage of participants = 36, 95% CI [27 to 44] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Combined Darbepoetin Alfa 300 μg; Test type: Superiority or Other; Percentage of participants = 38, 95% CI [29 to 47] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

8. Secondary Outcome: Number of Participants With ≥ 1 Red Blood Cell Transfusion From Week 1 to End of Study, by IV Iron Usage
Description: as for outcome 7
Time Frame: From Week 1 to Week 16
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 122 | 116
Participants | 47 | 41
Statistical Analysis 1: Comparison: Combined With Iron Groups; Test type: Superiority or Other; Percentage of participants = 35, 95% CI [27 to 44] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Combined Without Iron Groups; Test type: Superiority or Other; Percentage of participants = 39, 95% CI [30 to 47] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

9. Secondary Outcome: Number of Participants With ≥ 1 Red Blood Cell Transfusion From Week 5 to End of Study
Description: Number of participants with ≥ 1 RBC transfusion from Week 5 to end of study (Week 16)). Participants with a hemoglobin value ≤ 8 g/dL but no RBC transfusion were counted as having had a transfusion.
Time Frame: From Week 5 to Week 16
Population: Subset of Primary Analysis Set, composed of all randomized participants who received at least one dose of blinded study medication, and who were eligible for an RBC transfusion at week 5.
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa 300 μg Plus Iron | Darbepoetin Alfa 300 μg | Darbepoetin Alfa 500 μg Plus Iron | Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 56 | 60 | 59 | 57
Participants | 14 | 17 | 18 | 15
Statistical Analysis 1: Comparison: Darbepoetin Alfa 500 μg; Test type: Superiority or Other; Percentage of participants = 26, 95% CI [15 to 38] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Darbepoetin Alfa 500 μg Plus Iron; Test type: Superiority or Other; Percentage of participants = 31, 95% CI [19 to 42] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 3: Comparison: Darbepoetin Alfa 300 μg; Test type: Superiority or Other; Percentage of participants = 28, 95% CI [17 to 40] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 4: Comparison: Darbepoetin Alfa 300 μg Plus Iron; Test type: Superiority or Other; Percentage of participants = 25, 95% CI [14 to 36] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

10. Secondary Outcome: Number of Participants With a Hematopoietic Response, by Darbepoetin Alfa Dose
Description: Number of participants with a hematopoietic response, defined as > 2 g/dL increase from baseline or hemoglobin ≥ 12 g/dL during the treatment period in the absence of a red blood cell transfusion within the prior 28 days.
Time Frame: From Week 1 to Week 16
Population: Subset of Primary Analysis Set, composed of all participants who were randomized, properly consented, and received at least one dose of blinded study drug, who had a baseline hemoglobin value.
Measure: Number; unit: Participants
Arm/Group | Combined Darbepoetin Alfa 300 μg | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 118 | 120
Participants | 70 | 81
Statistical Analysis 1: Comparison: Combined Darbepoetin Alfa 500 μg; Test type: Superiority or Other; Percentage of participants = 68, 95% CI [59 to 76] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Combined Darbepoetin Alfa 300 μg; Test type: Superiority or Other; Percentage of participants = 59, 95% CI [50 to 68] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

11. Secondary Outcome: Number of Participants With a Hematopoietic Response, by IV Iron Usage
Description: Number of participants with a hematopoietic response, defined as > 2 g/dL increase from baseline or hemoglobin ≥ 12 g/dL during the treatment period in the absence of a red blood cell transfusion within the prior 28 days. Assessing the effect of iron in a factorial experiment.
Time Frame: From Week 1 to Week 16
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 122 | 116
Participants | 65 | 86
Statistical Analysis 1: Comparison: Combined Without Iron Groups; Test type: Superiority or Other; Percentage of participants = 53, 95% CI [44 to 62] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages
Statistical Analysis 2: Comparison: Combined With Iron Groups; Test type: Superiority or Other; Percentage of participants = 74, 95% CI [66 to 82] — Binomial proportion with confidence limit calculation using the normal approximation, and converted to percentages

12. Secondary Outcome: Time to Hematopoietic Response, by Darbepoetin Alfa Dose
Description: The time to hematopoietic response is the interval in weeks between study day 1 and the first day that a hematopoietic response is observed during the treatment period. Hematopoietic response is defined as an increase in hemoglobin concentration of ≥ 2.0 g/dL from baseline or a hemoglobin concentration ≥ 12.0 g/dL in the absence of RBC transfusions on the day of measurement and during the preceding 28 days of the treatment period. If a participant did not achieve a hematopoietic response by the time of withdrawal or the end of the treatment period (EOTP), the time to hematopoietic response was censored on the day of the last hemoglobin measurement or the EOTP, whichever was earlier. Median was calculated using using Kaplan-Meier estimates.
Time Frame: From Week 1 to Week 16
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Combined Darbepoetin Alfa 300: Darbepoetin alfa 300 μg subcutaneous injection with or without intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
Arm/Group | Combined Darbepoetin Alfa 300 | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 118 | 120
Weeks | 11.0 [8.0 to 12.0] | 9.0 [8.0 to 10.0]

13. Secondary Outcome: Time to Hematopoietic Response, by IV Iron Usage
Description: as for outcome 12
Time Frame: From Week 1 to Week 16
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 122 | 116
Weeks | 12.0 [10.0 to 15.0] | 8.0 [7.0 to 9.0]

14. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy (FACT) - Fatigue Score, by Darbepoetin Alfa Dose
Description: Health related quality of life was measured using the Functional Assessment of Cancer Therapy (FACT) - Fatigue subscale. The FACT-F includes 13 fatigue items, with each item assessed on a 5-point scale (ie, response values of 0 to 4). The FACT-F subscale score ranges from 0 to 52, where a higher score represents less fatigue.
Time Frame: Baseline and Week 16
Population: Patient-Reported Outcomes (PRO) Analysis Set, composed of all participants who were randomized, properly consented, and received at least one dose of blinded study drug, and who completed at least one baseline and one post-baseline PRO assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combined Darbepoetin Alfa 300 μg | Combined Darbepoetin Alfa 500 μg
Number analyzed (Participants) | 114 | 114
Units on a scale | 3.1 (11.8) | 0.6 (12.5)

15. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy (FACT) - Fatigue Score, by IV Iron Usage
Description: as for outcome 14
Time Frame: Baseline and Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combined Without Iron Groups | Combined With Iron Groups
Number analyzed (Participants) | 115 | 113
Units on a scale | 1.0 (13.1) | 2.7 (11.2)

ADVERSE EVENTS:
Time Frame: From first dose date to 3 weeks after the last dose of study drug or IV iron (Week 16).
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. One patient who was randomized to the 300 μg without iron arm received commercial iron product and was counted in the 300 μg with iron arm.
Groups:
- Darbepoetin Alfa 300 µg (Without IV Iron): Darbepoetin alfa 300 μg subcutaneous injection every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
- Darbepoetin Alfa 300 µg Plus Iron: Darbepoetin alfa 300 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
- Darbepoetin Alfa 500 µg (Without Iron): Darbepoetin alfa 500 μg subcutaneous injection every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
- Darbepoetin Alfa 500 µg Plus Iron: Darbepoetin alfa 500 μg subcutaneous injection plus intravenous (IV) iron 400 mg, every three weeks (Q3W), for up to 15 weeks (a total of 5 doses).
Arm/Group | Darbepoetin Alfa 300 µg (Without IV Iron) | Darbepoetin Alfa 300 µg Plus Iron | Darbepoetin Alfa 500 µg (Without Iron) | Darbepoetin Alfa 500 µg Plus Iron
Serious Adverse Events (participants affected / at risk) | 26/61 | 18/57 | 19/60 | 23/60
Other Adverse Events (participants affected / at risk) | 48/61 | 46/57 | 51/60 | 48/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa 300 µg (Without IV Iron) (N=61) | Darbepoetin Alfa 300 µg Plus Iron (N=57) | Darbepoetin Alfa 500 µg (Without Iron) (N=60) | Darbepoetin Alfa 500 µg Plus Iron (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 5 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enlarged uvula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Asthenia (General disorders) | 2 | 2 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 1 | 0
Disease progression (General disorders) | 2 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 3 | 5
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 4 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 1 | 3 | 2
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa 300 µg (Without IV Iron) (N=61) | Darbepoetin Alfa 300 µg Plus Iron (N=57) | Darbepoetin Alfa 500 µg (Without Iron) (N=60) | Darbepoetin Alfa 500 µg Plus Iron (N=60)
Anaemia (Blood and lymphatic system disorders) | 12 | 12 | 14 | 9
Leukopenia (Blood and lymphatic system disorders) | 9 | 7 | 6 | 9
Neutropenia (Blood and lymphatic system disorders) | 9 | 5 | 6 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 11 | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 7 | 3 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 5 | 3
Constipation (Gastrointestinal disorders) | 6 | 4 | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 6 | 11 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 4 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 13 | 5 | 10 | 11
Vomiting (Gastrointestinal disorders) | 10 | 3 | 3 | 6
Asthenia (General disorders) | 6 | 6 | 6 | 6
Disease progression (General disorders) | 1 | 5 | 1 | 4
Fatigue (General disorders) | 27 | 17 | 20 | 19
Mucosal inflammation (General disorders) | 3 | 3 | 0 | 1
Oedema peripheral (General disorders) | 9 | 4 | 7 | 6
Pain (General disorders) | 4 | 3 | 8 | 1
Pyrexia (General disorders) | 3 | 3 | 4 | 2
Urinary tract infection (Infections and infestations) | 4 | 2 | 3 | 1
Weight decreased (Investigations) | 3 | 2 | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 7 | 6 | 9 | 4
Decreased appetite (Metabolism and nutrition disorders) | 7 | 5 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 4 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 2
Dizziness (Nervous system disorders) | 4 | 3 | 7 | 7
Neuropathy (Nervous system disorders) | 2 | 1 | 2 | 5
Insomnia (Psychiatric disorders) | 6 | 5 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 6 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 2
Hypotension (Vascular disorders) | 4 | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.